CLINICAL TRIAL: NCT05639335
Title: Effects of Characters on Parents' Perceptions of Breakfast Cereals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-3135
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Character Control (Other): Participants will view images of three breakfast cereals (Frosted Flakes, Apple Jacks, Froot Loops) containing no characters.
  Interventions: Other: No Character Control
- Character (Experimental): Participants will view images of three breakfast cereals (Frosted Flakes, Apple Jacks, Froot Loops) containing their respective brand characters (e.g., Tony the Tiger) and a licensed character recently featured on these cereal brands (e.g., Buzz Lightyear).
  Interventions: Other: Experimental Characters

INTERVENTIONS:
Other: No Character Control — Participants will view images of three breakfast cereals (Frosted Flakes, Apple Jacks, Froot Loops) containing no characters.
  Arms: No Character Control
Other: Experimental Characters — Participants will view images of three breakfast cereals (Frosted Flakes, Apple Jacks, Froot Loops) containing their respective brand characters (e.g., Tony the Tiger) and a licensed character recently featured on these cereal brands (e.g., Buzz Lightyear).
  Arms: Character

SUMMARY:
Purpose: To test how the presence of characters on breakfast cereals affects parents' perceptions and purchase intentions for their children.

Participants: ~1,000 parents of children ages 2-12 Procedures: After completing a screener and reviewing a consent form, participants will complete two unrelated experimental studies. Participants will then move on to this study, where they will be randomized into conditions and view three breakfast cereal box images, with or without characters. They will then be asked a series of questions about their children and their perceptions about the breakfast cereals

DETAILED DESCRIPTION:
The use of characters, such as cartoons, is a prolific form of child-oriented marketing and may have particularly persuasive power in children. Parents and caregivers - who make most food purchases for children - are also persuaded by child-oriented marketing practices. The purpose of this study is to examine the impact of characters on parents' perceptions and purchase intentions of a breakfast cereal product.

Setting: This is an online study using Qualtrics. Recruitment: Participants will be recruited by Qualtrics panel company, a survey research firm through which participants are recruited voluntarily.

Informed Consent: Participants will read a written consent document that includes information about the study's purpose, expectations, and possible risks and benefits. Participants will acknowledge that they have read and agreed to the terms by clicking forward.

Randomization: Participants will be randomly assigned to one of two groups: 1.) control (breakfast cereal boxes with no characters) or 2.) characters (breakfast cereal boxes with a brand and at least one licensed character). Participants will view three brands (Frosted Flakes, Apple Jacks, Froot Loops).

Assessment: Using an online platform (Qualtrics), participants will complete an eligibility screener prior to the first experiment. They will then complete two unrelated experimental studies before beginning the current study. Participants will then be randomized into a condition and shown an image of the three cereal brands in random order. After each brand exposure, participants will be asked to respond to a series of questions measuring the following constructs: purchase intentions, perceived healthfulness, and perceived child appeal. After viewing all three brands and answering the aforementioned questions, participants will be queried on their perceptions of their child's perceived food-fussiness. Demographic information, such as age, gender, race/ethnicity, education, and income will be gathered at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Parent or guardian of at least one child between the ages of 2-12

Exclusion Criteria:

* <18 years old
* is not the parent or guardian of a child between the ages of 2-12

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1017 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Purchase intentions | During ~15 minute online survey
  The primary outcome will be purchase intentions, measured using the following item: "How likely would you be to buy this cereal to your [age]-year-old child in the next month?" using a 5-point likert-style response scale ranging from "not at all likely" (1) to "extremely likely" (5).

SECONDARY OUTCOMES:
Perceived healthfulness | During ~15 minute online survey
  Perceived healthfulness will be measured using the following item: "How healthy or unhealthy would it be for your [age] year old child to eat this cereal every day?" with a 5-point likert-style response scale ranging from "very unhealthy"(1) to "very healthy."(5)
Perceived child appeal | During ~15 minute online survey
  Perceived child appeal will be measured using three items adapted from previous research.
  Item 1: "How much do you think your child would enjoy eating this cereal?" (5-point likert scale, ranging from "not at all" (1) to "a great deal" (5)) Item 2: "How much do you think your [age]-year-old child would like the taste of this cereal?" (5-point likert scale, ranging from "not at all" (1) to "a great deal" (5)) Item 3: "How much do you think your [age]-year-old child would want to eat this cereal?" (5-point likert scale, ranging from "not at all" (1) to "a great deal" (5))

OTHER OUTCOMES:
Past week cereal consumption | During ~15 minute online survey
  Participants will be asked to report their child's past-week breakfast cereal consumption with the following question: "In the past week, how many days did your [age]-year-old child eat cereal?" (Measured using drop down menu, ranging from 0-7 days).
Perceived child food fussiness | During ~15 minute online survey
  Perceived child food fussiness will be assessed with a subset of the Food Fussiness Subscale. The following items will be queried:
  Item 1: My [piped age]-year-old child is interested in tasting food they haven't tasted before. (5-point likert scale, ranging from never (1) to always (5)) Item 2: My child [piped age]-year-old child decides that they don't like a food, even without tasting it. (5-point likert scale, ranging from never (1) to always (5)) Item 3: My [piped age]-year-old child enjoys tasting new foods.(5-point likert scale, ranging from never (1) to always (5)) Item 4: My [piped age]-year-old child refuses to eat new foods at first.(5-point likert scale, ranging from never (1) to always (5)).

CONTACTS AND LOCATIONS:
Overall Officials: Marissa G Hall, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset and analysis syntax that underlie the publication of the main study findings will be uploaded to a public website upon publication of the paper.
Supporting Information: SAP, Analytic Code
Time Frame: Within 6 months of publication
Access Criteria: No access criteria, will be publicly available. We plan to make these resources available on Open Science Framework.

REFERENCES:
- [Background] Hall MG, Lazard AJ, Grummon AH, Mendel JR, Taillie LS. The impact of front-of-package claims, fruit images, and health warnings on consumers' perceptions of sugar-sweetened fruit drinks: Three randomized experiments. Prev Med. 2020 Mar;132:105998. doi: 10.1016/j.ypmed.2020.105998. Epub 2020 Jan 23. PMID 31982477
- [Background] Liem DG, Zandstra LH. Children's liking and wanting of snack products: Influence of shape and flavour. Int J Behav Nutr Phys Act. 2009 Jul 2;6:38. doi: 10.1186/1479-5868-6-38. PMID 19573228
- [Background] Dial LA, Musher-Eizenman DR. Power of packaging: Evaluations of packaged fruits and vegetables by school-age children in the U.S. Appetite. 2020 May 1;148:104591. doi: 10.1016/j.appet.2020.104591. Epub 2020 Jan 9. PMID 31927069
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591